CLINICAL TRIAL: NCT00459043
Title: Randomized Phase II Study of Docetaxel in Combination With Zactima (ZD6474) in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Docetaxel in Combination With Zactima (ZD6474) in Patients With Locally Advanced Squamous Cell Carcinoma of the the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Loyola University (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Medical Oncology, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-283
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — vandetanib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Docetaxel Alone
  Interventions: Drug: Docetaxel
- 2 (Active Comparator): Docetaxel with ZD6474
  Interventions: Drug: ZD6474; Drug: Docetaxel

INTERVENTIONS:
Drug: ZD6474 — Taken orally once every morning
  Other Names: Zactima
  Arms: 2
Drug: Docetaxel — Given on the first day of every treatment cycle (every 3 weeks)

SUMMARY:
In this research study, the researchers are comparing the combination of docetaxel and Zactima with docetaxel alone to see if the combination of the two drugs will be more effective than docetaxel alone. Zactima blocks the actions of three substances in the body: 1)vascular endothelial growth factor reception (VEGFR); 2)epidermal growth factor receptor (EGFR); and 3) rearranged during transfection (RET). VEGFR stimulates the growth of new blood vessels. When certain proteins bind to the VEGF receptor, a process begins to occur which allows new blood vessels to be made that provide blood to the cancer cells. Zactima is thought to block these proteins from binding to the VEGF receptor, which would then block the process that creates new blood vessels. EGFR controls how quickly cells grow and multiply. RET is thought to have a particularly significant role in the development and growth of squamous cell tumors. The actions of Zactima are very different from the way standard chemotherapy drugs work. Researchers believe that Zactima might have different side effects from other cancer treatments so another one of the purposes of this study is to assess the side effects caused by the drug.

DETAILED DESCRIPTION:
* Participants will be "randomized" into one of the following study groups: Docetaxel or Docetaxel with Zactima. Randomization means that participants will be put into a group by chance.
* The Docetaxel group will receive docetaxel on the first day of every treatment cycle, which lasts for 3 weeks. Even though treatment will occur once every three weeks, participants will return to the clinic on a weekly basis for the first two cycles. After the first two cycles, they will only have to return to the clinic at the start of each cycle.
* The combination Docetaxel and Zactima group will also receive docetaxel once every three weeks. In addition to the docetaxel, they will also take a Zactima pill orally every morning. They will also have to return to the clinic on a weekly basis just as those in the docetaxel only group.
* The following tests and procedures will be performed during each cycle of treatment, regardless of which group the participant is randomized into. These are considered standard of care for treating patients with chemotherapy for recurrent head and neck cancer: physical exams; blood tests; urine test; nasopharyngoscopy; repeat imaging of the tumor (x-ray, CT, MRI or PET); photographs of the tumor. In addition to the tests mentioned above, the Zactima group will have EKGs performed 3 times on the first day of treatment, once at week 2, then at the beginning of cycles 2 and 3, and then every 6 weeks.
* Participants will continue on the study as long as they are receiving benefit and are not experiencing any unmanageable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically documented SCCHN, excluding nasopharyngeal carcinoma. Squamous cell carcinomas of unknown primary are allowed. Primary salivary gland tumors and tumor of the nasal cavity and paranasal sinuses are not included.
* 18 years of age or older.
* Evaluable or uni-dimensionally measurable local-regional and/or metastatic disease that is not amendable to primary surgical resection or radiotherapy.
* Life expectancy of at least 3 months.
* ECOG performance status of 0-2.
* Negative pregnancy test for women of childbearing potential.
* Adequate bone marrow function.

Exclusion Criteria:

* Evidence of sever or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the trial.
* Clinically significant cardiac event such as myocardial infarction, NYHA classification of heart disease grade II or higher within 3 months of study entry, or presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
* History of arrhythmia which is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
* Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication.
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age.
* Presence of left bundle branch block.
* QTc with Bazett's correction that is unmeasurable or > 480 msec on screening ECG.
* Any concomitant medication that may cause QTC prolongation, induce Torsades de Pointes or induce CYP3A4 function.
* Hypertension not controlled by medical therapy.
* Currently active diarrhea that may affect the ability of the patient to absorb Zactima.
* Pregnant or breast-feeding women.
* Previous or concurrent malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in-situ and adequately treated basal cell or squamous cell carcinoma of the skin.
* Receipt of any investigational agents within 30 days prior to commencing study treatment.
* Prior treatment with docetaxel.
* Last dose of prior chemotherapy discontinued less than 3 weeks before start of study therapy.
* Last dose of radiation therapy within the last 4 weeks before the start of study therapy, except palliative radiotherapy.
* Major surgery within 4 weeks, or incompletely healed surgical incision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Loyola University Medical Center/Cardinal Bernadin Cancer Center, Maywood, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2007 to October 2009, 30 patients were enrolled from four different sites in United States.
Pre-assignment Details: Patients were randomized in a 1:1 ratio to receive docetaxel alone or docetaxel and vandetanib as combination therapy. No stratification at randomization was made for the study
Groups:
- 1Docetaxel Single Agent: Docetaxel 75 mg/m2 was administered every 21 days intravenously.
- 2 Combination Docetaxel and ZD6474: Docetaxel with ZD6474
  Docetaxel 75 mg/m2 was administered every 21 days intravenously. ZD6474 (Vandetanib) at 100 mg was administered as a once daily tablet given orally.
Period: Overall Study
Arm/Group | 1Docetaxel Single Agent | 2 Combination Docetaxel and ZD6474
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: One patient withdrew consent after being randomized to docetaxel alone arm and did not receive any treatment, therefore, 29 patients were analyzable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel Single Agent | Combination of Docetaxel and Zactima | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 4 | 4 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (42) | 60 (35) | 58 (46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 10 | 14 | 24
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Partial Response Rate in Both Groups of Patients.
Description: Objective tumor response was evaluated radiogically using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. For target lesions: Complete Response (CR) disappearance of all target lesions; Partial Response (PR) >= 30% decrease in the sum of the longest diamter of target lesions; Overall Response (OR) = CR+PR
Time Frame: 3 years
Population: 29 patients were analyzable
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 1Docetaxel Single Agent: Docetaxel Alone
- 2 Combination Docetaxel and ZD6474: Docetaxel with ZD6474
Arm/Group | 1Docetaxel Single Agent | 2 Combination Docetaxel and ZD6474
Number analyzed (Participants) | 14 | 15
percentage of participants | 7 [0.2 to 33.8] | 13 [1.6 to 40.4]

2. Secondary Outcome: Progression Free Survival
Description: Progression is defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as a 20% increase in the sumof the longest diameter of target lesions, or a measurable increase in a non-target lesion or the appearance of new lesions
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 1Docetaxel Single Agent | 2 Combination Docetaxel and ZD6474
Number analyzed (Participants) | 14 | 15
weeks | 3.21 [3.0 to 22.0] | 9 [5.86 to 18.1]

3. Secondary Outcome: Overall Survival
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 1Docetaxel Single Agent | 2 Combination Docetaxel and ZD6474
Number analyzed (Participants) | 14 | 15
weeks | 26.8 [17.7 to 100.7] | 24.1 [16.4 to 171.1]

ADVERSE EVENTS:
Arm/Group | 1Docetaxel Single Agent | 2 Combination Docetaxel and ZD6474
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/15
Other Adverse Events (participants affected / at risk) | 14/14 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1Docetaxel Single Agent (N=14) | 2 Combination Docetaxel and ZD6474 (N=15)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1Docetaxel Single Agent (N=14) | 2 Combination Docetaxel and ZD6474 (N=15)
Neutrophils (Blood and lymphatic system disorders) | 11 | 10
Dysphagia (Gastrointestinal disorders) | 8 | 8
Constipation (Gastrointestinal disorders) | 6 | 7
Diarrhea (Gastrointestinal disorders) | 2 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 7
Hemoglobin (Blood and lymphatic system disorders) | 4 | 7
Neutrophils (Blood and lymphatic system disorders) | 7 | 6
Hemorrhage (Blood and lymphatic system disorders) | 1 | 6
Mucositis/Stomatitis (Gastrointestinal disorders) | 4 | 5
Anorexia (Gastrointestinal disorders) | 2 | 5
Pain (General disorders) | 5 | 2
Depression (Psychiatric disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes